CLINICAL TRIAL: NCT02583035
Title: Telephone OncoGériatric Followed in the Management of Elderly Patients Treated for Cancer or Haematological Malignancy
Acronym: TelOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TelOG
Record Dates: First submitted 2015-09-17; First posted 2015-10-21 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Cancer; Hematologic Malignancy
Keywords: cancer; geriatric
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nurse telephone contact (Other): 3 days of consultation, telephone follow-up of the patient by the nurse coordinator of the Geriatric Oncology Unit to validate
  Interventions: Other: Nurse telephone contact

INTERVENTIONS:
Other: Nurse telephone contact — Nurse will contact patient 3 days before consultation

SUMMARY:
There are no recommendations and few studies on the monitoring of fragile patients in the oncological treatment, both on the organizational arrangements on its interest in the prevention of functional deterioration of the patient and adaptation of the potential cancer treatment.

The oncogériatrique evaluation being time-consuming, requiring the movement of these more or less frail elderly patients, it seems difficult to envisage repeated and systematic standardized geriatric assessments during cancer treatment. Geriatric fragility can be detected by telephone. Craven et al. has already assessed the telephone follow-up by a nurse in patients treated for cancer, but with the aim to detect toxicities of cancer treatment, patients are not very old (mean age 64.8 years).

External evaluation by the nurse coordinator of UCOG (Coordination Unit in geriatric oncology) not knowing the patients included avoids bias of subjectivity in the interrogation.

However the telephone monitoring, with the aim to evaluate the evolution of geriatric frailty, has not been specifically studied in the elderly population treated for cancer, while taking oncology load.

The investigators wish to study the feasibility and validity of telephone follow-up which could eventually be used routinely to identify patients requiring further medical consultation oncogériatrique.

ELIGIBILITY:
Inclusion Criteria:

* Patients 70 years and older with cancer or hematologic malignancies;
* Faced benefit from cancer treatment (systemic treatment, curative radiotherapy) in one of the clinical sites;
* Addressed in onco-gériatric consultation in the usual routine care sector;
* Mastery of the French language;
* Patient affiliated to the social security system;
* Patient has given its written consent.

Exclusion Criteria:

* Life expectancy <3 months
* Inability to communicate by telephone (deafness, speech disorder, ..)
* Inability collection of written consent
* Group 4 SiO (International Society of Geriatric Oncology), Performance status (PS) 4
* initial MMSE (Mini-Mental State Examination) <18/30
* oncological treatment envisaged: analgesic radiotherapy or exclusive decompressive, brain radiation therapy in toto
* Patient under guardianship

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 131 (Actual)
Dates: Start 2015-02; Primary Completion 2018-02-16 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
Memory on the Mini Mental Scale | 3 months after inclusion
Falls on the number of falls | 3 months after inclusion
Pain on the EVS (verbal scale) scale | 3 months after inclusion
Autonomy on the ADL (activities of daily living) score | 3 months after inclusion
Pain on the EN (numericale scale) scale | 3 months after inclusion
Autonomy on the IADL (The Lawton Instrumental Activities of Daily Living Scale ) score | 3 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Bérengère Beauplet, MD, Principal Investigator — University Hospital, Caen
Locations (5):
- France (5):
  - Centre Hospitalier, Bayeux
  - CHU, Caen
  - Centre François Baclesse, Caen
  - Centre Hospitalier, Dieppe
  - Centre Hospitalier du Havre, Le Havre